CLINICAL TRIAL: NCT06470659
Title: Effectiveness of a Telehealth Medical Weight Management Program Prescribing Anti-obesity Medications Paired With a Digital Behavioral Weight Management Program
Brief Title: Medications With or Without WeightWatchers
Acronym: Meds WOW-WW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Cardel, PhD, MS, RD (Industry)
Responsible Party: Sponsor-Investigator, Michelle Cardel, PhD, MS, RD, Senior Director of Global Clinical Research and Nutrition, WW International Inc
Organization: WW International Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Meds WOW-WW
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meds alone (No Intervention): Participants in this group do not receive behavioral or lifestyle support alongside their medications. The medications are not part of the intervention (it is part of the eligibility criteria).
- Meds plus WW (Experimental): Participants in this group receive behavioral or lifestyle support from WW Clinic alongside their medications. The medications are not part of the intervention (it is part of the eligibility criteria).
  Interventions: Behavioral: WW Clinic

INTERVENTIONS:
Behavioral: WW Clinic — Telehealth platform that specializes in medical weight management and integrates the behavioral and lifestyle support from WW
  Arms: Meds plus WW

SUMMARY:
The study compares the effectiveness of adults living with overweight or obesity taking weight management medications alone vs taking them with behavioral and lifestyle support. The primary outcome is percent body weight lost at 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI of >30 or BMI of >27 with one or more weight related medically qualifying condition (hypertension, dyslipidemia, sleep apnea, cardiovascular disease)
* Determined eligible for Bupropion/Naltrexone or Liraglutide by WW Clinic medical provider and initiated a medication management plan

Exclusion Criteria:

* Diabetes
* Uncontrolled hypertension
* History of seizures
* History of glaucoma
* History of chronic kidney disease
* Currently taking bupropion
* Currently taking naltrexone
* Current or previous history of anorexia or bulimia nervosa
* Engagement with vomiting or laxative use within the last 28 days with the aim of controlling their shape or weight
* Currently taking opioids
* Previous surgical obesity treatment
* Use of other anti-obesity medication in last 90 days or a GLP1 in the last 180 days
* Lost weight >11 lbs in the last 90 days
* Pregnant, breastfeeding, intends to become pregnant, of child-bearing potential and not using a highly effective contraceptive method
* Any other reason rendering a participant unsuitable for trial participation, as determined by a clinician or study investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Percent body weight lost at 12 weeks | Baseline, 12 weeks
  Measurement of weight using a bluetooth body weight scale

SECONDARY OUTCOMES:
Change in body weight (in kg or pounds) at 12 weeks | Baseline, 12 weeks
  Measurement of weight using a bluetooth body weight scale
Physical Activity and Sedentary Behavior | Baseline, 12 weeks
  The Global Physical Activity Questionnaire (GPAQ) is a 16 item scale.
Dietary Intake | Baseline, 12 weeks
  Diet ID is powered by Diet Quality Photo Navigation (DQPN®). It is a digital toolkit and 1 component will be used in the study: ID assessment.
Habit/Automaticity | Baseline, 12 weeks
  The Self-Report Behavioral Automaticity Index (SRBAI) is a 4-item measure.
Hunger VAS (Visual Analogue Scale) | Baseline, 12 weeks
  The Hunger VAS (Visual Analogue Scale) is a reliable measure for appetite research. The Hunger VAS asks "How hungry did you feel over the past week" and is composed of a line with words anchored at each end describing the extremes (Not at all hungry, Extremely hungry). Participants are asked to make a mark on the line corresponding to their feelings and quantification of the measurement is done by measuring the distance from the left end of the mark.
Impact on Quality of Life | Baseline, 12 weeks
  The Impact of Weight on Quality of Life-Lite (IWQOL-Lite) is a validated self-report measure for an individual's perception of how their weight affects their day-to-day life
Well-being | Baseline, 12 weeks
  The World Health Organization (WHO-5) Well-being Index consists of five statements, which respondents rate, in relation to the past two weeks, using a six-point Likert scale
Body Appreciation | Baseline, 12 weeks
  The Body Appreciation Scale (BAS-2) measures individuals acceptance of, favorable opinions toward, and respect for their bodies. There are 10 items, each assessed on a scale from 1-never to 5-always. Higher scores indicate higher body appreciation.
Food Cravings | Baseline, 12 weeks
  The Food Cravings Inventory (FCI-II) is a 33-item self-report measure designed to assess the subjective experience of food craving across 33 different foods
Self-Compassion | Baseline, 12 weeks
  The Self-Compassion Scale (SCS) is a 26-item measure of self-compassion that is psychometrically valid and theoretically coherent. The SCS consists of six subscales:
  self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identified.
  Subscales are computed by calculating the mean of subscale item responses. A total self-compassion score can be obtained by reverse scoring the negative subscale items (self-judgment, isolation, and over-identification) and computing a grand mean of all six subscale means. Higher scores indicate greater self compassion.
Weight Bias | Baseline, 12 weeks
  The Weight Bias Internalization Scale (WBIS-2F) has 13 items and responses are rated on a 7-point Likert scale(strongly disagree -strongly agree). Responses provide insight on the participant's internalized beliefs and feelings regarding their weight. There are two subscales: Weight-Related Distress (7 items; 7-13; Cronbach's alpha =0.910) and Weight-Related Self-Devaluation (6 items; 1-6; Cronbach's alpha =0.763). The WBIS-2F has been tested for validity in people with overweight and obesity and the two factor model demonstrated good to excellent fit with the data. Scores are calculated by taking an average of the response values. Questions 1,2,4,5, should be reverse scored before calculating the average. Higher scores indicating greater internalized weight bias.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Cardel, PhD, RD, Principal Investigator — WW International Inc; Rebecca Jones, PhD, Principal Investigator — WW International Inc
Locations (1):
- WW International, Inc, New York, New York, United States